Rituximab for Schizophrenia Spectrum Disorder. A Pilot Study.

NCT03983018 Unique Protocol ID: EudraCT Number: 2018-004618-17

Study Title: Rituximab - Immunotherapy for Schizophrenia spectrum disorder in adults. An open pilot study.

Protocol Number: RITS-PS-2019 EudraCT Number: 2018-004618-17

Protocol Date: 2019-01-28 Protocol Version: 1.2

Informed consent final version 21st of May 2019

## Rituximab for Schizophrenia Spectrum Disorder. A Pilot Study.

## NCT03983018 Unique Protocol ID: EudraCT Number: 2018-004618-17

## **Consent to Participate in the Study**

I have received oral and written information about the study and have had the opportunity to ask questions. I may keep the written information.

| | | YES NO |
|---|---|---|
| <ul> <li>I consent to participate in the stress</li> <li>Spectrum Disorder. A Pilot Stud</li> </ul> | | |
| which means that: | | |
| | v information being processed in the manner descripant information. | ribed in the |
| - | samples being stored in a biobank in the manner pant information. | described in the |
| c. I consent to the | study monitor accessing medical records for data | a verification. |
| I consent to providing a cerebros | pinal fluid sample via lumbar puncture. | |
| I consent to undergoing an MRI | scan. | |
| I consent to providing a stool san | mple. | |
| I consent to undergoing an intest | inal examination (with biopsy). | |
| Place | Date | |
| Participant's signature | Printed name | |
| Responsible researcher | Printed name | |